CLINICAL TRIAL: NCT00464425
Title: Electroacupuncture for Postoperative Ileus After Laparoscopic Colorectal Surgery: a Randomised Sham-controlled Pilot Study
Brief Title: Electroacupuncture for Postoperative Ileus After Laparoscopic Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Simon SM Ng, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2006.429-T
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Postoperative Ileus
Keywords: Electroacupuncture; Postoperative ileus; Colorectal surgery; Laparoscopic surgery; Randomised trial
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electroacupuncture (EA) (Experimental): EA using sharp needles placed at various acupoints; electrical stimulation at 50 Hz applied to the needles
  Interventions: Procedure: Electroacupuncture
- Sham Acupuncture (SA) (Sham Comparator): Acupuncture using blunt-tip needles placed 15 mm away from acupoints; no electrical stimulation used
  Interventions: Procedure: Sham Acupuncture
- No Acupuncture (NA) (No Intervention): Control
  Interventions: Other: No Acupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — EA using sharp needles placed at various acupoints; electrical stimulation at 50 Hz applied to the needles
  Other Names: EA
  Arms: Electroacupuncture (EA)
Procedure: Sham Acupuncture — Acupuncture using blunt-tip needles placed 15 mm away from acupoints; no electrical stimulation used
  Other Names: SA
  Arms: Sham Acupuncture (SA)
Other: No Acupuncture — Control
  Arms: No Acupuncture (NA)

SUMMARY:
Postoperative ileus remains a significant medical problem after colorectal surgery that adversely influences patients' recovery and prolongs hospital stay. In fact, a substantial portion of the overall hospitalisation period after colorectal surgery is attributed to the time it takes for ileus to resolve. Although laparoscopic colorectal surgery has been proven to be associated with better short-term clinical outcomes including faster return of gastrointestinal function than open surgery, the duration of postoperative ileus in the laparoscopic arm is still reported to be as long as 4 days in most of the randomised trials. Additional measures are thus necessary to further enhance the gastrointestinal recovery after laparoscopic colorectal surgery in order to maximise its benefits, and acupuncture may be one of the options. Acupuncture is widely accepted in China as well as throughout the world as an effective treatment option for the management of postoperative nausea and vomiting and various functional gastrointestinal disorders. Its role in treating postoperative ileus, however, is less clear, and data from the Chinese as well as the Western literature are scarce. We therefore propose to carry out a prospective randomised sham-controlled pilot study to assess the efficacy of electroacupuncture in treating postoperative ileus after laparoscopic colorectal surgery. The acupoints relevant to the treatment of abdominal distension and constipation, including Zusanli (stomach meridian ST-36), Sanyinjiao (spleen meridian SP-6), Hegu (large intestine meridian LI-4), and Zhigou (triple energizer meridian TE-6) will be used.

DETAILED DESCRIPTION:
Postoperative ileus remains a significant medical problem after colorectal surgery that adversely influences patients' recovery and prolongs hospital stay. In fact, a substantial portion of the overall hospitalisation period after colorectal surgery is attributed to the time it takes for ileus to resolve. Different treatment modalities including thoracic epidural analgesia, pharmacological therapy, early enteral feeding, and early mobilisation have been attempted, but none has an established role as a specific remedy for postoperative ileus. Although laparoscopic colorectal surgery has been proven to be associated with better short-term clinical outcomes including faster return of gastrointestinal function than open surgery, the duration of postoperative ileus in the laparoscopic arm is still reported to be as long as 4 days (which is just about 1 day earlier than that in the open arm) in most of the randomised trials. Additional measures are thus necessary to further enhance the gastrointestinal recovery after laparoscopic colorectal surgery in order to maximise its benefits, and acupuncture may be one of the options. Acupuncture is widely accepted in China as well as throughout the world as an effective treatment option for the management of postoperative nausea and vomiting and various functional gastrointestinal disorders. Its role in treating postoperative ileus, however, is less clear, and data from the Chinese as well as the Western literature are scarce. Besides, the heterogeneity of the study designs and flaws in methodology of the reported studies have made interpretation of these data difficult. Results of the present study can provide evidence-based clarification of the role of acupuncture in treating postoperative ileus after laparoscopic colorectal surgery. If the hypothesis is proven to be correct and substantiated by further studies, the incorporation of electroacupuncture into any fast-track recovery programmes after laparoscopic, open, or even emergency colorectal surgery should be considered. As laparoscopic colorectal surgery has been shown to have higher direct cost than the open counterpart, a faster postoperative recovery may help to reduce the financial burden to the hospital and improve the cost-effectiveness of the procedure.

Patients will be enrolled into the study if all the inclusion and exclusion criteria are satisfied after the laparoscopic surgery. Randomisation will be done shortly after surgery. Patients will be randomised to receive either electroacupuncture (EA group), sham acupuncture (SA group), or no acupuncture (NA group). The medical acupuncturist is the only individual who is aware of the treatment allocation; patients of the EA and SA groups are blinded to the treatment. The patients randomised to the EA and SA groups will undergo 1 session of acupuncture daily from postoperative day 1 till day 4. Adverse events associated with acupuncture including bleeding, dizziness, excessive pain, and allergic reaction will be closely monitored. The acupuncture needle will be immediately withdrawn if these events occur.

The postoperative management of all patients will be standardised. Pethidine 1mg/kg as postoperative analgesia will be given every 4-hourly on demand. Early ambulation will be encouraged. Oral feeding will be resumed as soon as gastrointestinal function returns clinically (no nausea or vomiting, no abdominal distension, passage of flatus or stool). No gum chewing will be allowed. Patients will be discharged when they tolerate diet and are fully ambulatory.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients undergoing elective laparoscopic resection of colonic and upper rectal cancer without the need of conversion
2. Patients with American Society of Anaesthesiologists grading I-III
3. Informed consent available

Exclusion Criteria:

1. Patients undergoing laparoscopic low anterior resection with total mesorectal excision, abdominoperineal resection, and total/proctocolectomy
2. Patients undergoing simultaneous laparoscopic resection of colorectal cancer and other coexisting intraabdominal diseases (e.g. liver metastasis, symptomatic gallstones)
3. Patients undergoing laparoscopic resection of colorectal cancer with en-bloc resection of surrounding organs (e.g. small bowel, urinary bladder)
4. Patients who developed intraoperative problems or complications (e.g. bleeding, tumour perforation) that required conversion
5. Patients with intestinal obstruction
6. Patients with previous history of abdominal surgery
7. Patients with stoma creation
8. Patients with evidence of peritoneal carcinomatosis
9. Patients who are expected to receive epidural opioids for postoperative pain management
10. Patients who are allergic to acupuncture needles

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Time to defaecation, measured in days, from the time the laparoscopic surgery ends till the first observed passage of stool | Up to 1 month

SECONDARY OUTCOMES:
Time of first passing flatus reported by the patients (days) | Up to 1 month
Time to resume normal diet (days) | Up to 1 month
Time to walk independently (days) | Up to 1 month
Duration of hospital stay (days) | Up to 1 month
Pain scores on visual analogue scale (from 0 which implies no pain at all, to 10 which implies the worst pain imaginable) on the first 3 postoperative days | Up to 1 month
Postoperative analgesic requirement (number of doses on 50-mg Pethidine). | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, FRCSEd (Gen), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Surgical Wards 4C and 4D, Prince of Wales Hospital, Shatin, Hong Kong SAR, China

REFERENCES:
- [Derived] Ng SSM, Leung WW, Mak TWC, Hon SSF, Li JCM, Wong CYN, Tsoi KKF, Lee JFY. Electroacupuncture reduces duration of postoperative ileus after laparoscopic surgery for colorectal cancer. Gastroenterology. 2013 Feb;144(2):307-313.e1. doi: 10.1053/j.gastro.2012.10.050. Epub 2012 Nov 6. PMID 23142625